CLINICAL TRIAL: NCT03738137
Title: Narcotrend Versus Bispectral Index Monitoring During Sufentanil-Midazolam Anesthesia for Bronchoscopy Under Conscious Sedation
Brief Title: Narcotrend Versus Bispectral Index Monitoring During Sufentanil-Midazolam Anesthesia for Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Professor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NTBIS2018
Record Dates: First submitted 2018-11-01; First posted 2018-11-13 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Bronchoscopy
Keywords: Narcotrend; Bispectral index; Bronchoscopy; Conscious Sedation
MeSH Terms: interventions — Sufentanil; Lidocaine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Narcotrend (Experimental): After 0.1µg/kg sufentanil is applied, miidazolam is given by non-anaesthetist physicians to achieve moderate levels of sedation as assessed by the Narcotrend index stage C.
  Interventions: Device: Narotrend; Drug: Sufentanil; Drug: Lidocaine; Drug: Midazolam
- BIS (Experimental): After 0.1µg/kg sufentanil is applied, midazolam is given by non-anaesthetist physicians to achieve moderate levels of sedation as assessed by bispectral index (BIS; between 70 and 85).
  Interventions: Device: BIS; Drug: Sufentanil; Drug: Lidocaine; Drug: Midazolam
- No monitoring (Experimental): After 0.1µg/kg sufentanil is applied, midazolam iss given by non-anaesthetist physicians according to patient's tolerance .
  Interventions: Drug: Sufentanil; Drug: Lidocaine; Drug: Midazolam
- Lidocaine (Experimental): Only topical anesthesia was applied.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Device: Narotrend — Narcotrend motoring
  Arms: Narcotrend
Device: BIS — Bispectral index monitoring
  Arms: BIS
Drug: Sufentanil — sufentanil is applied.
  Arms: BIS; Narcotrend; No monitoring
Drug: Lidocaine — Topical Anesthesia
Drug: Midazolam — midazolam is applied.
  Arms: BIS; Narcotrend; No monitoring

SUMMARY:
This study was aimed to determine whether narcotrend monitoring was better than bispectral index monitoring during sufentanil-midazolam anesthesia for bronchoscopy under conscious sedation. Patients were randomised to receive Narcotrend, Bispectral Index(BIS) monitoring or without monitoring. Midazolam was given by non-anaesthetist physicians to achieve moderate levels of sedation as assessed by the narcotrend index (NI; B and C) or bispectral index (BIS; between 70 and 85) or according to patient's tolerance assessed by physician . The primary end-point was dosage of midazolam. Other end-points included adverse events, patient tolerance and physician satisfaction.

ELIGIBILITY:
Inclusion Criteria:

ASA grade I-II

Exclusion Criteria:

1. psychological disorders
2. SpO2<90% in ambient air
3. hypersensitivity or allergy to anaesthetic drugs or benzodiazepine
4. severe chronic obstructive pulmonary disease (forced expiratory volume in 1 s ,50% of predicted value, requirement for oxygen therapy)
5. unstable haemodynamic status
6. habitual alcohol consumption

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Dosage of Midazoam | during the procedure
  dosage of midazolam

SECONDARY OUTCOMES:
patient's subjective tolerance | 30minutes after bronchoscopy
  the intensity of four key symptoms during bronchoscopy (pain, nausea, breathlessness and cough) and memory using a visual analogic scale (VAS: 1 mm: excellent tolerance, 100 mm very low tolerance)
patient's global tolerance assessed by operator | 30minutes after bronchoscopy
  the global tolerance of patient to the procedure using a visual analogic scale (VAS: 1 mm: excellent tolerance, 100 mm very low tolerance)
adverse events rate | every 3 minutes during the procedure and at 5, 15 and 30 minutes thereafter.
  hypotension (systolic BP <100 mmHg or mean arterial blood pressure (MAP)<60 mmHg), tachycardia (fC>100/min and/or a variation of >20% from baseline value), oxygen desaturation (SaO2 decrease<90% for >30 s), bradycardia (HR<50/min).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China